CLINICAL TRIAL: NCT05252338
Title: A Phase 1, Open-label, Dose-escalation, First-in-human, Clinical Trial to Evaluate the Safety, Reactogenicity and Immunogenicity of the Investigational Seasonal Quadrivalent Influenza mRNA Vaccine CVSQIV Administered Intramuscularly in Healthy Younger and Older Adults
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Vaccine CVSQIV in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CV-SQIV-001
Record Dates: First submitted 2022-01-26; First posted 2022-02-23 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Safety; Reactogenicity; Immunogenicity; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Younger Adults group aged 18-55 years (Experimental): Subjects will be enrolled in a staggered manner in up to 5 dose levels (provisional dose levels of 3, 6, 12, 20 and 28µg). All subjects will receive a single dose of CVSQIV on Day 1.
  Interventions: Biological: CVSQIV
- Adults group aged ≥65 years (Experimental): Subjects will be enrolled in a staggered manner in up to 5 dose levels (provisional dose levels of 3, 6, 12, 20 and 28µg). All subjects will receive a single dose of CVSQIV on Day 1.
  Interventions: Biological: CVSQIV

INTERVENTIONS:
Biological: CVSQIV — Participants will receive an intramuscular injection by needle in the deltoid area.

SUMMARY:
This study aims to evaluate the safety and reactogenicity profile of CVSQIV at different dose levels.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose-escalation FIH trial to evaluate the safety, reactogenicity and immunogenicity of different dose levels of CVSQIV using an adaptive dose-finding design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 18 and 55 years, inclusive, at enrollment (Younger Adults groups) or aged ≥65 years at enrollment (Older Adults groups). A healthy subject is defined as an individual who is in good general health, according to the Investigator's assessment. Chronic health conditions are acceptable if the condition is considered stable and well controlled with treatment according to the discretion of the Investigator.
* Signed informed consent obtained before any trial procedures.
* Expected to be compliant with protocol procedures and available for clinical follow-up through the last planned contact.
* Physical examination without clinically significant findings according to the Investigator's assessment.
* Body mass index (BMI) ≥18.0 and ≤32.0kg/m2.
* Females: At the time of enrollment, negative human chorionic gonadotropin (hCG) pregnancy test (serum) for women presumed to be of childbearing potential on the day of enrollment. On Day 1 (pre-vaccination): negative urine pregnancy test (hCG), (only required if serum pregnancy test was performed more than 3 days before). Note: Women that are postmenopausal (defined as amenorrhea for ≥12 consecutive months prior to enrollment without an alternative medical cause) or permanently sterilized will be considered as not having reproductive potential.
* Females of childbearing potential must use highly effective methods of birth control from 1 month before until 3 months after the trial vaccine administration. The following methods of birth control are considered highly effective when used consistently and correctly:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable);
  * Intrauterine devices;
  * Intrauterine hormone-releasing systems;
  * Bilateral tubal occlusion;
  * Vasectomized partner;
  * Same sex relationships.

Sexual abstinence (periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal) are not acceptable methods.

Exclusion Criteria:

* Use of any investigational or non-registered product (vaccine or drug) other than the trial vaccine within 28 days preceding the trial vaccine administration, or planned use during the trial.
* Receipt of any influenza vaccine within 90 days of enrollment.
* Receipt of any mRNA vaccine within 2 months of enrollment.
* Receipt of any other vaccines within 28 days prior to enrollment or planned receipt of any vaccine within 28 days of trial vaccine administration.
* Any treatment with immunosuppressants or other immune-modifying drugs (including, but not limited to, corticosteroids, biologicals and methotrexate) for >14 days total within 6 months prior to the trial vaccine administration or planned use during the trial, with the exception of inhaled or topically-applied steroids. For corticosteroid use, this means prednisone or equivalent, 0.5 mg/kg/day for 14 days or more.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination, including known human immunodeficiency virus infection.
* Chronic hepatitis B virus infection and chronic hepatitis C virus infection.
* History of pIMD
* History of angioedema.
* History of any neurological disorders or seizures including Guillain-Barré syndrome, with the exception of febrile seizures during childhood.
* History of allergy to any component of CVSQIV, or to aminoglycoside or beta-lactam antibiotics.
* History of any severe allergic reaction or anaphylactic reaction.
* History of or current alcohol and/or drug abuse.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the trial vaccine administration.
* Presence or evidence of significant acute or chronic medical or psychiatric illness.
* Current or past malignancy, unless completely resolved without sequelae for >5 years.
* For females: pregnancy or lactation.
* Subjects with impaired coagulation or any bleeding disorder in whom an intramuscular injection or a blood draw is contraindicated.
* Subjects employed by the Sponsor, Investigator or trial site, or relatives of research staff working on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
The frequencies of Grade 3 ARs and any SAR within at least 20 hours after the trial vaccine administration by dose level, for decisions on subsequent vaccination of additional sentinel subjects with the same dose level. | up to day 2
The frequencies of Grade 3 ARs and any SAR within at least 60 hours after the trial vaccine administration by dose level, for decisions on dose escalation as well as continuation of enrollment at the same dose level. | up to day 3
The frequencies, intensities and duration of solicited local ARs on the day of vaccination and the following 7 days by dose level, for the characterization of the safety and reactogenicity profile. | up to day 8
The frequencies, intensities, duration and relationship to trial vaccination of solicited systemic AEs on the day of vaccination and the following 7 days by dose level, for the characterization of the safety and reactogenicity profile. | up to day 8
The occurrence, intensities and relationship to trial vaccination of unsolicited AEs on the day of vaccination and the following 28 days by dose level, for the characterization of the safety and reactogenicity profile. | up to day 29
The occurrence and relationship to trial vaccination of SAEs and AESIs throughout the trial, for the characterization of the safety and reactogenicity profile. | through study completion, an average of 6 months

SECONDARY OUTCOMES:
For each antigen, the proportion of subjects with antigen-specific serum HAI assay titers. | On Day 22 and Day 183
For each antigen, geometric mean titers (GMTs) of antigen-specific HAI antibody titers. | On Day 22 and Day 183
For each antigen, the proportion of subjects with antigen-specific seroconversion measured by HAI assay. | On Day 22 and Day 183
For each antigen, the percentage of subjects with a post-vaccination HAI antibody titer ≥1:20, ≥1:40 and ≥1:80. | On Day 22 and Day 183

CONTACTS AND LOCATIONS:
Locations (3):
- Panama (3):
  - International Vaccination and Research Center (CEVAXIN) Avenida Mexico, 33 Street, Panama City, Calidonia, Panama City
  - International Vaccination and Research Center (CEVAXIN) Panama Clinic, Ramon H Jurado Street, Pacific Center, Level 12, Panama City
  - Unidad de Investigación Clínica INDICASAT AIP / Hospital Paitilla, Panama City